CLINICAL TRIAL: NCT06652945
Title: Efficacy of Uterine Artery Embolization (UAE) in Management of Symptomatic Uterine Adenomyosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Gamal Hassan, Assistant Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uterine Artery Embolization
Record Dates: First submitted 2024-10-15; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Uterine Adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — Uterine Artery Embolization; Polyvinyl Alcohol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Symptomatic uterine adenomyosis (Experimental): Patients with symptomatic uterine adenomyosis
  Interventions: Other: Uterine artery embolization

INTERVENTIONS:
Other: Uterine artery embolization — Uterine artery embolization under fluoroscopy
  Other Names: Fluoroscopy; polyvinyl alcohol (PVA)

SUMMARY:
Aim of the work:

Evaluating the efficiency of uterine artery embolization as a minimally invasive method of treatment in management of symptomatic women with uterine adenomyosis

DETAILED DESCRIPTION:
Adenomyosis is defined as a non-neoplastic disease, caused by benign invasion of the myometrial layer by endometrial tissue, associated with myometrial smooth muscle hyperplasia. This ectopic endometrium shows two main patterns of distribution in the myometrium: either focal endometrial implant of endometrial glands, or diffuse invasion of the myometrium. Uterine enlargement is often seen with diffuse adenomyosis, while in cases with focal adenomyosis, characteristic feature in ultrasound (US) can be misdiagnosed as leiomyoma, appearing as focal heterogeneous myometrial thickening or myometrial cysts.

Usually, adenomyosis is presented with dysmenorrhea, menorrhagia, and abnormal uterine bleeding. Previously, adenomyosis was diagnosed in multiparous women older than 40 years, causing abnormal uterine bleeding (AUB). But recently, it has been widely recognized among larger group, including nulliparous women earlier in reproductive life, owing to increased availability and better imaging techniques.

The first imaging modality to diagnose adenomyosis is transabdominal sonography (TAS) or transvaginal sonography (TVS). While magnetic resonance (MR) imaging is considered the gold standard diagnosis method due to its accuracy; being noninvasive modality and its ability for better soft tissue characterization to differentiate adenomyosis from other pathologies.

First line of management of adenomyosis include medications as non-steroidal anti-inflammatory drugs and/or hormonal therapy. Yet, other methods of treatment are needed in different cases.

For many years, the most common line of treatment for symptomatic uterine adenomyosis is hysterectomy. Some studies discussed the possibility of uterine-sparing surgeries to treat adenomyosis, despite the controversy of application. Many patients prefer uterine-sparing lines of treatment over hysterectomy, especially after failure of medical treatment. Recent studies have been investigating uterine artery embolization (UAE) as a promising line of treatment of adenomyosis.

In 1995, the study of Ravina was the first to discuss UAE. Ever since, UAE was established as a treatment option for symptomatic patients with adenomyosis, as well as uterine fibroids, owing to its earliest positive results. The objective of UAE is to produce more than 34% necrosis of adenomyotic tissues, using trans-arterial catheters. Recent studies show increasing success rates of managing adenomyosis using UAE, with rates ranging from 60% to 70% and from 72% to 94.3%, respectively.

To evaluate uterine volume and areas of necrosis, patients are referred to perform MRI following the UAE, as in cases with fibroid disease. With regard of different symptoms and presentations of adenomyosis, having a cut-off value to evaluate effectiveness of the procedure to alleviate the symptoms is considered challenging.

Some major complications and side effects can occur such as infections, and pain caused by ischemic necrosis, especially the first hours after the procedure which require strong regimen for pain control. Six percent of the cases complained of persistent amenorrhea, and they were above the age of 40 years old.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* Symptomatic pure adenomyosis or dominant adenomyosis when both adenomyosis and fibroids coexist
* Women with an indication for hysterectomy (either failed or refused medical treatment).

Exclusion Criteria:

* Patients under 18 years of age,
* Patients with pelvic infection,
* Suspected or confirmed malignancy
* Current or future desire to conceive
* Deep infiltrating endometriosis requiring surgery or obstructing the bowel, or
* Coexisting hysteroscopically removable submucous fibroids
* Any absolute contraindication to angiography such as:
* hypersensitivity to intravenous contrast media,
* impaired coagulation profile or
* impaired renal function.

Ages: 35 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Management of symptomatic uterine adenomyosis | three years
  Relieving the symptoms of uterine adenomyosis using uterine artery embolization such as abnormal uterine bleeding and dysmenorrhea

IPD SHARING:
Plan to Share IPD: Yes